CLINICAL TRIAL: NCT00002352
Title: Pilot Study of the Antiviral Activity of Multiple Doses of Oral Lobucavir in AIDS Patients
Brief Title: A Study of Lobucavir in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 248A; AI459-007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — lobucavir

INTERVENTIONS:
Drug: Lobucavir

SUMMARY:
The purpose of this study is to see if lobucavir is a safe and effective treatment for cytomegalovirus in patients with AIDS.

DETAILED DESCRIPTION:
Patients receive 1 of 2 doses of lobucavir for 28 days, with 2 weeks of follow-up. Weekly clinic visits are required.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine.
* TMP / SMX.
* Isoniazid.
* Dapsone.
* Fluconazole.
* Ketoconazole.
* Rifabutin.
* Fluoxetine HCl.
* Acetaminophen.
* Antacids.
* Metamucil.
* Multivitamins.
* Other drugs with approval from sponsor.

Patients must have:

* AIDS.
* CD4 count < 200 cells/mm3.
* Cytomegalovirus ( CMV ) viruria and virosemenia.
* No evidence of intraocular CMV.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Acute or chronic cardiovascular, pulmonary, renal, hepatic, pancreatic, hematologic, endocrine, neurological, or other unstable illness.
* Inability to take oral medication.
* Allergy to nucleoside analogs.
* Diarrheal illness.
* Poor venous access.
* Positive test for drugs of abuse.
* Any other condition that would render patient unsuitable for study.

Patients with the following prior conditions are excluded:

* History of pancreatitis.
* Recent diarrheal illness.
* History of weight loss.
* Acute serious illness within 4 weeks prior to study entry.

Prior Medication:

Excluded within 4 weeks prior to study entry:

* Erythropoietin.
* Any agent with anti-CMV activity.
* Other investigational agents.

Prior Treatment:

Excluded within 4 weeks prior to study entry:

* Surgery.
* Blood transfusion. Drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - San Francisco Veterans Adm Med Cntr, San Francisco, California
  - Univ of Minnesota, Minneapolis, Minnesota